CLINICAL TRIAL: NCT04289038
Title: Evaluation of the Efficacy of VR and AR on Pruritus Symptoms in Patients Receiving Hemodialysis Treatment
Brief Title: The Efficacy of VR and AR on Pruritus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Baskent University (Other)
Responsible Party: Principal Investigator, Neşe Altinok Ersoy, MS, Research Assistant, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KA180157
Record Dates: First submitted 2020-01-16; First posted 2020-02-28 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Chronic Renal Insufficiency; Pruritus; Itch
Keywords: itch; pruritus; nursing; virtual reality
MeSH Terms: conditions — Renal Insufficiency, Chronic; Pruritus | interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Autogenic Relaxation (Experimental): Autogenic Relaxation: It is an exercise program consisting of standard sentences that describe the body's absolute comfort and calm features.
  Interventions: Other: Autogenic Relaxation
- Virtual Reality (Experimental): Virtual reality: Playing games via smart phone with virtual reality glasses and headset.
  Interventions: Other: virtual reality game application
- Control Group (Other): Routine nursing care and kidney function narration
  Interventions: Other: kidney function narration

INTERVENTIONS:
Other: Autogenic Relaxation — Autogenic relaxation
  Arms: Autogenic Relaxation
Other: virtual reality game application — virtual reality game application,
  Arms: Virtual Reality
Other: kidney function narration — kidney function narration
  Arms: Control Group

SUMMARY:
The research will be conducted randomly in order to determine the effect of VR and AR on pruritus symptom.

DETAILED DESCRIPTION:
In this study, there will be three groups: intervention group 1 with autogenic relaxation (AR), intervention group 2 with virtual reality (VR) game application and control group with routine nursing care and kidney functions narration. The number of volunteers to be included in the study was determined by power analysis. Forty patients with itch symptoms will be included in each group. Preliminary application for all three groups will be performed in the patient group registered to the Dialysis Unit of the Nephrology Department of Hacettepe University and Baskent University Hospital. Socio-Demographic Form, 5-D Itch Scale, Dermatology Life Quality Index, State and Trait Anxiety Scale, Pruritus Behavior and SGO / OR Application Log.

ELIGIBILITY:
Inclusion Criteria:

* Receiving hemodialysis treatment for the last 6 months,
* Receiving four hour hemodialysis treatment three times a week,
* 18-65 years of age,
* experiencing pruritus for the last month.
* Not taking any pharmacological / non-pharmacological treatment for pruritus
* No cognitive and psychiatric diagnosis,
* Do not use hearing aids,
* Open to communication and cooperation,
* Using smart mobile phone,
* Without liver disease and dermatological diseases,
* Patients who agree to participate in the study will be included in the study.

Exclusion Criteria:

* Pregnant in the research process,
* Kidney transplantation,
* Experiencing discomfort due to virtual reality glasses,
* Patients who voluntarily leave the trial will be excluded from the follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2022-02-26 (Actual)

PRIMARY OUTCOMES:
5-D Itch Scale | Assessing change of 5-D Itch Scale scores baseline, first, fifth and seventh weeks.
  The score obtained from information about itching severity, frequency, and its effect on daily life activities.

SECONDARY OUTCOMES:
Dermatology Life Quality Index | Assessing change of Dermatology Life Quality Index scores baseline, first, fifth and seventh weeks. .
  The scale gives an information about quality of life
State-Trait Anxiety Inventory | Assessing change of State-Trait Anxiety Inventory scores baseline, first, fifth and seventh weeks.
  The scale gives an information about anxiety

CONTACTS AND LOCATIONS:
Overall Officials: NEŞE ALTINOK ERSOY, PHDC, Principal Investigator — Hacettepe University
Locations (1):
- Neşe Altinok Ersoy, Ankara, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Altinok Ersoy N, Akyar I, Yildirim T, Erdogmus S. Effects of a Virtual Reality Game or Autogenic Relaxation on Pruritus, Anxiety and Dermatologic Quality of Life in Haemodialysis Patients: A Randomized Controlled Trial. Int J Nurs Pract. 2025 Oct;31(5):e70071. doi: 10.1111/ijn.70071. PMID 41069201